CLINICAL TRIAL: NCT07203859
Title: Comparison of the Effects of Ultrasound-Guided Quadro-İliac Plane Block on Postoperative Pain Level and Analgesia Requirement in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: The Effectiveness of Quadro İliac Plane Block in Percutaneous Nephrolithotomies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2025-07/32
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Percutaneous Nephrolithotomy
Keywords: postoperative pain; regional anesthesia; percutaneous nephrolithotomy; quadroiliac plane block; opioid free analgesia; ibuprofen; novel fascial plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No non-routine procedures will be performed on this group.
- Quadro-İliac Plane Block(QİPB) (Active Comparator): For this group, after the surgical procedure is completed, the patient will be placed in a lateral position with the operated side facing up, and a QIPB will be performed. With the patient in the lateral position, the spinous process of the L3 vertebra will first be imaged with an ultrasound probe positioned transversely in the midline. Then, by slightly shifting the probe laterally, the transverse process of the vertebra will be visualized within the erector spinae muscle. The probe will then be rotated in the sagittal plane and advanced caudally about 1 cm, visualizing the crista iliaca. On the cranial side of the crista iliaca, the erector spinae muscle, quadratus lumborum, and psoas major muscles will be visualized sequentially. With the needle direction cranial to caudal, the crista iliaca will be gently touched, and the needle will be positioned between the erector spinae and the quadratus lumborum muscle. After injecting 40 ml of 0.25% bupivacaine, the needle will be injected.
  Interventions: Procedure: Quadro-İliac Plane Block(QİPB)

INTERVENTIONS:
Procedure: Quadro-İliac Plane Block(QİPB) — 40 mL of 0.25% bupivacaine
  Arms: Quadro-İliac Plane Block(QİPB)

SUMMARY:
Our aim was to investigate the effect of quadro iliac plane block on postoperative analgesia in patients undergoing percutaneous nephrolithotomy surgery and to determine which areas of the skin this block anesthetizes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who underwent percutaneous nephrolithotomy under general anesthesia and were I-II-III according to the American Society of Anesthesiologists (ASA) risk classification were included in the study.

Exclusion Criteria:

* patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with known allergies to any of the study drugs,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment
* patients who wanted to withdraw from the study,
* patients with alcohol and drug addiction,
* patients with musculoskeletal abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Scores | Postoperative 24 hours
  Description: Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Dermatome Area | Postoperative 2 hours
Total tramadol consumption | Postoperative 24 hours
  Postoperative total analgesic need was recorded as "milligram" in unit.

CONTACTS AND LOCATIONS:
Overall Officials: OĞUZ GÜNDOĞDU, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation; SAMET YENİHAN, Study Chair — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No